CLINICAL TRIAL: NCT06629766
Title: The EPIC Study: Exploring Paternal Age and the Influence on Blastocyst Culture
Acronym: EPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2405-BRG-141-KB
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Infertility (IVF Patients); Oocyte Competence; Sperm DNA Fragmentation; Paternal Age; Sperm Selection
Keywords: microfluidic; density grade centrifugation; sperm selection; paternal age; sperm DNA fragmentation; Zymot
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oocytes inseminated by sperm prepared by a microfluidic (Zymot) sperm preparation device (Experimental): Half of the mature oocytes will be randomly allocated to receive sperm prepared by the microfluidic (Zymot) sperm preparation device. This sperm will be used by the embryologist for the ICSI procedure.
  Interventions: Device: Microfluidic sperm separation device
- Oocytes inseminated by sperm prepared via density grade centrifugation (Other): The other half of the mature oocytes will be allocated to receive sperm prepared by DGC. This sperm will be used by the embryologist for the ICSI procedure.
  Interventions: Other: Density grade centrifugation

INTERVENTIONS:
Device: Microfluidic sperm separation device — An aliquot of 850ul will be used for the Zymot sperm selection device. The sperm processing via Zymot will be per manufacturer's guidelines
  Other Names: Zymot
  Arms: Oocytes inseminated by sperm prepared by a microfluidic (Zymot) sperm preparation device
Other: Density grade centrifugation — 5ul of the ejaculated sample will be assessed for DGC via Makler assessment. If the sample for DGC is adequate per lab standard operating procedures, then routine DGC sperm preparation and embryologist sperm selection for the ICSI procedure will occur.
  Arms: Oocytes inseminated by sperm prepared via density grade centrifugation

SUMMARY:
This study aims to assess the effect of age of the male partner and the reproductive ability of sperm prepared via sperm selection devices (Zymot) compared to routine embryologist selected sperm after density gradient centrifugation (DGC) preparation for intracytoplasmic sperm injection (ICSI) in patients undergoing in vitro fertilization treatment (IVF) of their infertility.

DETAILED DESCRIPTION:
In this study, we aim to determine the clinical utility of the Zymot sperm selection methodology for ICSI, while also accounting for paternal age. This study will be a prospective, split cohort, randomized, control trial comparing the routine standard of DGC sperm preparation for ICSI versus sperm prepared via Zymot for ICSI. Embryology parameters, ploidy status, DNA fragmentation and clinical pregnancy outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing first IVF cycle
* Electing single embryo transfer
* Electing PGT-A of their embryos
* Female partners age <42 years old at start of VOR cycle, but >18 years old.
* AMH ≥ 1.2 ng/mL
* AFC ≥ 8
* FSH ≤ 12IU/L
* At least 4 mature oocytes (M2s) retrieved at the VOR procedure in order to randomize
* Intention to transfer the morphological best quality, euploid, embryo at the frozen embryo transfer procedure

Exclusion Criteria:

* Contraindication to IVF
* Clinical indication for preimplantation genetic testing (i.e., screening for single gene disorder, chromosomal translocation, or any other disorders requiring a more detailed embryo genetic analysis)
* Male partner with azoospermia or oligozoospermia (<500,000 total motile spermatozoa on the most recent semen analysis within one year of enrollment)
* Planned for previously cryopreserved sperm to be used for ICSI
* Donor sperm
* Male partner with Y-chromosome microdeletion
* Male partner with any Karyotype other than 46,XY
* Male partner requiring surgically obtained sperm either via testicular or epididymal retrieval procedures
* Uncorrected hydrosalpinges that communicate with the endometrial cavity
* Endometrial Insufficiency, as defined by a prior cycle with maximal endometrial thickness <6mm,), or persistent endometrial fluid
* Donor oocyte or embryo cycles
* Gestational carriers

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blastulation Rate per Mature Oocyte (M2) | approximately 1 week post oocyte retrieval procedure
  count of blastocyst stage embryos per M2 count

SECONDARY OUTCOMES:
Fertilization Rate | approximately 24 hours post oocyte retrieval procedure
  count of fertilized zygotes (2 pronuclei (2PN)) per M2 count
Blastulation Rate per 2PN | approximately 1 week post oocyte retrieval procedure
  count of blastocyst stage embryos per 2PN
Blastocyst Morphology using Modified Gardner Scale | approximately 1 week post oocyte retrieval procedure
  Morphology Grade at time of trophectoderm biopsy and vitrification. Expansion 1-6. Inner cell mass and trophectoderm graded A-D.
Ploidy rates | approximately 2 weeks post blastocyst trophectoderm biopsy
  Rates of whole chromosome negative and positive preimplantation genetic testing for aneuploidy (PGT-A) results per blastocyst
Ongoing pregnancy rate | 6 weeks post embryo transfer
  rate of ongoing pregnancy at 8-9 weeks gestational age when discharged to obstetrician
Pregnancy Loss Rates | 1 day to 7 months post positive beta human chorionic gonadotrophin
  a loss of pregnancy (either biochemical or clinical)
Live birth rate | approximately 7 months after discharge to obstetrician
  rate of live born infants
Sperm DNA Fragmentation | approximately 1-3 hours post intracytoplasmic sperm injection procedure
  Sperm DNA Fragmentation will be run on remnant samples
Positive beta human chorionic gonadotrophin (bhcg) | 7-10 days post embryo transfer
  positive pregnancy test with bhcg >5mUI/mL
Embryological Efficiency | same day as ICSI procedure
  Sperm prep time (Time from embryologist possession of sample to completion of prep procedure and ICSI start), benchtop time, ICSI procedural time
Embryology Questionnaire | upon primary outcome completion in approximately 18 months
  Gain perspectives from lab personnel related to likeability, ease of use and efficiency between the two devices

CONTACTS AND LOCATIONS:
Overall Officials: Kassie Bollig, MD, MSCE, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No